CLINICAL TRIAL: NCT03620539
Title: Effects of Sauna Bathing on Cerebrovascular Function in Middle-aged to Older Adults With Heart Disease
Brief Title: Sauna Bathing to Improve Vascular Health of Adults With Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Daniel Gagnon, Researcher, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ICM2017-2312
Record Dates: First submitted 2018-07-24; First posted 2018-08-08 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease
Keywords: flow-mediated dilation; sauna; vascular; heat
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants randomized to the control condition will be asked to maintain their normal daily habits.
- Sauna (Experimental): The sauna intervention will consist of 20 to 30 minute sauna bathing sessions within a dry Finnish sauna, performed 4 times per week.
  Interventions: Other: Lifestyle intervention

INTERVENTIONS:
Other: Lifestyle intervention — Sauna bathing
  Arms: Sauna

SUMMARY:
This study is a clinical trial that will determine if sauna bathing improves blood vessel health in adults aged 50-70 years with heart disease.

DETAILED DESCRIPTION:
Mounting evidence suggests that heat therapy may improve cardiovascular health. Recent analyses of a large cohort of middle-aged to older Finnish men have established that frequent sauna bathing is associated with a reduced risk of cardiovascular mortality, of developing dementia and Alzheimer's disease, and of developing hypertension. Given the observational nature of these relationships, it remains unknown if the beneficial effects of sauna bathing can be directly attributed to heat exposure.

The objective of this study is to test the primary hypothesis that 8 weeks of sauna bathing improves flow-mediated dilation, a measure of blood vessel health, in middle-aged to older adults (50-70 yrs) with stable coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. A history of angiographic coronary disease: ≥70% arterial diameter narrowing of at least one major epicardial coronary artery and/or prior coronary revascularization and/or documented prior acute coronary syndrome and/or perfusion defect during exercise testing or pharmacological stimulation
2. Stable medication doses (≥4 weeks) prior to enrolment
3. Body mass index <35 kg/m2

Exclusion Criteria:

1. Recent (<3 months) coronary artery disease-related hospitalization or change in angina pattern
2. Unstable angina
3. Ejection fraction <40% and/or clinical evidence of heart failure
4. Significant valvular heart disease
5. Uncontrolled hypertension (>180/110 mmHg)

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation | Change from baseline after 8 weeks
  Brachial artery flow-mediated dilation in response to 5 minutes of forearm occlusion

SECONDARY OUTCOMES:
Post-occlusion reactive hyperaemia (AUC) | Change from baseline after 8 weeks
  Vascular conductance area-under-the-curve during reactive hyperaemia induced by 5 minutes of forearm occlusion
Post-occlusion reactive hyperaemia (Peak) | Change from baseline after 8 weeks
  Peak vascular conductance during reactive hyperaemia induced by 5 minutes of forearm occlusion
Local skin heating-induced vasodilation | Change from baseline after 8 weeks
  Plateau of the cutaneous vascular conductance response during local heating of the skin to 39°C

OTHER OUTCOMES:
Blood pressure | Change from baseline after 8 weeks
  Systolic blood pressure at rest
Central arterial stiffness | Change from baseline after 8 weeks
  Carotid-femoral pulse wave velocity
Heart rate variability | Change from baseline after 8 weeks
  Resting levels of heart rate variability

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Prevention and Rehabilitation Centre of the Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Debray A, Gravel H, Garceau L, Bartlett AA, Chaseling GK, Barry H, Behzadi P, Ravanelli N, Iglesies-Grau J, Nigam A, Juneau M, Gagnon D. Finnish sauna bathing and vascular health of adults with coronary artery disease: a randomized controlled trial. J Appl Physiol (1985). 2023 Oct 1;135(4):795-804. doi: 10.1152/japplphysiol.00322.2023. Epub 2023 Aug 31. PMID 37650138